CLINICAL TRIAL: NCT05866744
Title: Effects of a Time-restricted Hypocaloric Mediterranean Diet in Patients with Non-alcoholic Fatty Liver Disease on Glucose Metabolism (CHRONO-NAFLD Project)
Brief Title: Effects of Time-restricted Hypocaloric Diet in Patients with NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Collaborators: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRBD40/27.04.2022 716/26-11-22
Record Dates: First submitted 2023-03-30; First posted 2023-05-19 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Time-Restricted Feeding; Mediterranean Diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early Time-Restricted Feeding Plus Hypocaloric Mediterranean Diet (Experimental): Early 14:10 time-restricted feeding plus hypocaloric Mediterranean diet
  Interventions: Other: Early Time-Restricted Feeding Plus Hypocaloric Mediterranean Diet
- Late Time-Restricted Feeding Plus Hypocaloric Mediterranean Diet (Experimental): Late 14:10 time-restricted feeding plus hypocaloric Mediterranean diet
  Interventions: Other: Late Time-Restricted Feeding Plus Hypocaloric Mediterranean Diet
- Hypocaloric Mediterranean Diet Without Time Restriction In Feeding (Active Comparator): Hypocaloric Mediterranean diet without time restriction in feeding
  Interventions: Other: Hypocaloric Mediterranean Diet Without Time Restriction In Feeding

INTERVENTIONS:
Other: Early Time-Restricted Feeding Plus Hypocaloric Mediterranean Diet — 18 patients with NAFLD will be asked to follow an early 14:10 (14 hours fasting and 10 hours feeding) time-restricted (eating between 08:00-18:00) and individualized Mediterranean diet plan with caloric restriction (energy deficit of 500 kcal/day) for 12 weeks
  Arms: Early Time-Restricted Feeding Plus Hypocaloric Mediterranean Diet
Other: Late Time-Restricted Feeding Plus Hypocaloric Mediterranean Diet — 18 patients with NAFLD will be asked to follow a late 14:10 (14 hours fasting and 10 hours feeding) time-restricted (eating between 12:00-22:00) and individualized Mediterranean diet plan with caloric restriction (energy deficit of 500 kcal/day) for 12 weeks
  Arms: Late Time-Restricted Feeding Plus Hypocaloric Mediterranean Diet
Other: Hypocaloric Mediterranean Diet Without Time Restriction In Feeding — 18 patients with NAFLD will be asked to follow an individualized Mediterranean diet plan with caloric restriction (energy deficit of 500 kcal/day) without time restriction in feeding (eating throughout the day) for 12 weeks
  Arms: Hypocaloric Mediterranean Diet Without Time Restriction In Feeding

SUMMARY:
The effects of a time-restricted hypocaloric Mediterranean type diet compared to a conventional hypocaloric Mediterranean type diet on blood glucose metabolism and liver steatosis in people with non-alcoholic fatty liver disease will be investigated.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effects of the time in which food intake is restricted (morning or evening hours or no restriction in time) on glucose metabolism and liver steatosis in the context of a hypocaloric diet plan in 54 patients with non-alcoholic fatty liver disease (NAFLD). The participants will be divided into 3 groups of 18 individuals each and will be randomly assigned to one of the 3 dietary interventions. In the first group (control group), participants will be given a weight loss program based on the principles of the Mediterranean Diet (energy deficit of 500 kcal/day with the aim of losing 0.5 kg per week) with the instruction to consume their meals throughout the day, without time restriction. In the second group (early eaters), individuals will be given a weight loss program based on the principles of the Mediterranean Diet (energy deficit of 500 kcal/day with the aim of losing 0.5 kg per week), and they will be asked to consume all of their meals within 10 hours (between 07:00-09:00 and 17:00-19:00) and refrain from consuming caloric foods and drinks for the remaining 14 hours. In the third group (late eaters), individuals will be given a weight loss program based on the principles of the Mediterranean Diet (energy deficit of 500 kcal/day with the aim of losing 0.5 kg per week), and they will be asked to consume all of their meals within 10 hours (between 11:00-13:00 and 21:00-23:00) and refrain from consuming caloric foods and drinks for the remaining 14 hours.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >25 kg/m2
* Liver steatosis with Magnetic Resonance Elastography (MRE)

Exclusion Criteria:

* Other chronic liver diseases
* Alcohol consumption >20 g/day (female) and >30 g/day (male)
* Medications that cause liver disease or secondary NAFLD (e.g. tamoxifen, corticosteroids, Methotrexate, tetracycline, estrogens, valproic acid)
* Changes in body weight ± 3 % in the last 3 months
* Patients following a hypocaloric diet program and/or time-restricted feeding and/or other intermittent fasting protocols
* Unstable glucose-lowering medications in the last 6 months
* Body weight lowering medications and/or history of bariatric surgery
* Statins and/ or other fat-reducing medications if not taken in steady dosage for at least 3 months
* Uncontrolled type 2 diabetes mellitus defined as HbA1c value > 9.0% or insulin depending type 1 and 2 diabetes mellitus
* Pregnancy
* Lactation
* Immunologic or inflammatory diseases
* Depression and other psychiatric diseases
* Patients working in shifts
* Cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose concentrations | 12 weeks
  Clinically significant change in blood glucose concentrations (mg/dL)

SECONDARY OUTCOMES:
Change in body weight | 12 weeks
  Clinically significant change in body weight (kg)
Change in blood insulin concentrations | 12 weeks
  Clinically significant change in blood insulin concentrations (μU/L)
Change in Controlled Attenuation Parameter (CAP) | 12 weeks
  Clinically significant change in CAP (dB/m)
Change in blood lipids levels | 12 weeks
  Clinically significant change in triglycerides (mg/dL), total cholesterol (mg/dL), low-density lipoprotein (mg/dL) and high-density lipoprotein (mg/dl)
Change in Chronic Liver Disease Questionnaire (CLDQ) | 12 weeks
  Clinically significant change in health status within individuals with NAFLD. The CLDQ includes 29 items in the following domains: abdominal symptoms, fatigue, systemic symptoms, activity, emotional function and worry. Overall CLDQ scores calculated for each domain range from 1 (most impaired) to 7 (minimum frequency of symptoms). The total score is calculated as the average score of the 29 items.

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Laiko General Hospital of Athens, Athens, Attica
  - Agricultural University of Athens, Athens, Attica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsitsou S, Bali T, Adamantou M, Saridaki A, Poulia KA, Karagiannakis DS, Papakonstantinou E, Cholongitas E. Effects of a 12-Week Mediterranean-Type Time-Restricted Feeding Protocol in Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease: A Randomised Controlled Trial-The 'CHRONO-NAFLD Project'. Aliment Pharmacol Ther. 2025 Apr;61(8):1290-1309. doi: 10.1111/apt.70044. Epub 2025 Feb 28. PMID 40017349